CLINICAL TRIAL: NCT02228083
Title: Occurrence of Heart Arrhythmia During Restorative Dental Procedure Under Local Anesthesia , in Heart Failure Pacients. A Double-blind Study
Brief Title: Dental Anesthesia in Heart Failure Patients
Acronym: DAHFP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: InsufCard
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: dental; epinephrine; local anesthetic; lidocaine; cardiac arrhythmias; procedure
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safety of dental anesthesia (Active Comparator): Application of local dental anesthesia with two cartridges (5,6 mL) of the lidocaine 2% with epinephrine 1:100.000 in heart failure patients in functional class III or IV.
  Interventions: Drug: Lidocaine with epinephrine
- Oral health profile (Other): An oral health profile of patients with heart failure will be described based in oral clinical examination.
  Interventions: Drug: Lidocaine with epinephrine

INTERVENTIONS:
Drug: Lidocaine with epinephrine — Lidocaine without vasoconstrictor , lidocaine with epinephrine 1:100,000

SUMMARY:
To investigate the occurrence of arrhythmias in dental treatment with local anesthetic.

DETAILED DESCRIPTION:
Heart failure is defined as the inability of the heart to offer blood supply required to meet metabolic demand of the tissues and thus exercise adequately its role as a pump. According to data collected from the single health system (DATASUS), approximately 6.4 million Brazilians have heart failure. This large contingent of patients will require multi-professional treatment, in particular, careful with dental health heart failure is regarded as the final common pathway of most cardiovascular diseases and, after installation of symptoms (mainly in the stages of functional class NYHA III and IV) have poor prognosis with average survival of 1.7 years 3.2 years for men and for women. Dental treatment often requires application of local anesthetic. The adrenaline, agent vasoconstrictor, is widely used in dental treatment and aims to extend the effect of local anesthetic. Specifically in people with heart failure, there shortcomings of evidence in the literature, the harmful effects of adrenaline 1:100,000 added to the local anaesthetic lidocaine. Among the potential complications, we can highlight: arrhythmias, systemic blood pressure elevation and elevation of heart rate. The main objective of this work will investigate the occurrence of arrhythmias by evaluating of electrocardiographic parameters. Our secondary objectives will be assessing: variations of blood pressure by ambulatory blood pressure monitoring, cardiac frequency and chest pain. We will study 70 patients between 18 and 75 years with a diagnosis of congestive heart failure functional class NYHA III and IV and restorative dental treatment indication. A random picture in double-blind study, patients are divided into two groups, one group receives as local anesthetic lidocaine 2% with adrenaline 1 in comparison with the second group that will receive 2% lidocaine with vasoconstrictor.

ELIGIBILITY:
Inclusion Criteria:

* any race,nationality,profession, single or married.
* class II , III or IV of New York heart Association ( NYHA)
* minimum 45% ventricular ejection fraction
* patient must be in a clinical treatment or hospital treatment
* patient must need dental restorative treatment , mandible or maxilla, due to caries or need for substitution of a inadequate dental filling.

Exclusion Criteria:

* patients with history of heart attack within less than three months
* acute myocardial infarction
* unstable angina
* significant ventricular dysfunction
* severe ventricular arrhythmia
* malignant hypertension
* neoplasms
* sepsis
* pregnancy
* allergy to lidocaine and epinephrine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Heart rate (bpm) | 24 hours
  The continuous electrocardiogram recording for a period of 24 hours will be obtained through the Holter monitor model Seer Ligth (GE), with three channels (seven-way) cable, installed a half hour before the dental procedure. The first analysis will be done automatically by the computer system, followed by visual and manual review at which supraventricular and ventricular premature heartbeats will be filtered accurately.
  Electrocardiographic variables are: heart rate maximum, minimum and mean HR, supraventricular extrasystole (VES) and ventricular (EV) FC. The program shall provide the record in HR per minute for 24 hours. The average individual will be calculated for the period studied, to then calculate the sample mean and groups LSA and LCA. The ESV and EV will be identified in tracing obtained every minute. Consider the valid values recorded HR and ischemic episodes; analyze the occurrence of EV and ESV occurring in number> 10 per hour in both groups, by study period.

CONTACTS AND LOCATIONS:
Overall Officials: Itamara LI Neves, PhD, Principal Investigator — Instituto do Coração do HCFMUSP; Edimar A Bocchi, Habilitation, Study Director — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo; Ricardo S Neves, PhD, Study Chair — Instituto do Coração do HCFMUSP; Sergio ET Quaresma, MS., Study Chair — Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Coração HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Mann DL. Mechanisms and models in heart failure: A combinatorial approach. Circulation. 1999 Aug 31;100(9):999-1008. doi: 10.1161/01.cir.100.9.999. No abstract available. PMID 10468532
- [Background] Palatini P, Frigo G, Bertolo O, Roman E, Da Corta R, Winnicki M. Validation of the A&D TM-2430 device for ambulatory blood pressure monitoring and evaluation of performance according to subjects' characteristics. Blood Press Monit. 1998 Aug;3(4):255-260. PMID 10212363
- [Background] Sivaneswaran S. The oral health of adults in NSW, 2004-06. N S W Public Health Bull. 2009 Mar-Apr;20(3-4):46-51. doi: 10.1071/NB08066. PMID 19401068
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Result] [Guidelines of the Brazilian Cardiology Society to the diagnosis and treatment of heart failure]. Arq Bras Cardiol. 1999 Feb;72 Suppl 1:1-30. No abstract available. Portuguese. PMID 10488571
- [Result] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202
- [Result] Hunt SA, Baker DW, Chin MH, Cinquegrani MP, Feldman AM, Francis GS, Ganiats TG, Goldstein S, Gregoratos G, Jessup ML, Noble RJ, Packer M, Silver MA, Stevenson LW, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Jacobs AK, Hiratzka LF, Russell RO, Smith SC Jr; American College of Cardiology/American Heart Association. ACC/AHA guidelines for the evaluation and management of chronic heart failure in the adult: executive summary. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to revise the 1995 Guidelines for the Evaluation and Management of Heart Failure). J Am Coll Cardiol. 2001 Dec;38(7):2101-13. doi: 10.1016/s0735-1097(01)01683-7. No abstract available. PMID 11738322
- [Result] Hempenstall PD, Campbell JP, Bajurnow AT, Reade PC, McGrath B, Harrison LC. Cardiovascular, biochemical, and hormonal responses to intravenous sedation with local analgesia versus general anesthesia in patients undergoing oral surgery. J Oral Maxillofac Surg. 1986 Jun;44(6):441-6. doi: 10.1016/s0278-2391(86)80008-8. PMID 3009759
- [Result] Brand HS, Gortzak RA, Abraham-Inpijn L. Anxiety and heart rate correlation prior to dental checkup. Int Dent J. 1995 Dec;45(6):347-51. PMID 8666460
- [Result] Hasse AL, Heng MK, Garrett NR. Blood pressure and electrocardiographic response to dental treatment with use of local anesthesia. J Am Dent Assoc. 1986 Oct;113(4):639-42. doi: 10.14219/jada.archive.1986.0245. PMID 2945853
- [Result] Hill CM, Mostafa P, Stuart AG, Thomas DW, Walker RV. ECG variations in patients pre- and post-local anaesthesia and analgesia. Br Dent J. 2009 Dec 19;207(12):E23. doi: 10.1038/sj.bdj.2009.978. Epub 2009 Nov 6. PMID 19893562
- [Result] Neves RS, Neves IL, Giorgi DM, Grupi CJ, Cesar LA, Hueb W, Grinberg M. Effects of epinephrine in local dental anesthesia in patients with coronary artery disease. Arq Bras Cardiol. 2007 May;88(5):545-51. doi: 10.1590/s0066-782x2007000500008. English, Portuguese. PMID 17589629
- [Result] Perusse R, Goulet JP, Turcotte JY. Contraindications to vasoconstrictors in dentistry: Part I. Cardiovascular diseases. Oral Surg Oral Med Oral Pathol. 1992 Nov;74(5):679-86. doi: 10.1016/0030-4220(92)90365-w. PMID 1437073
- [Result] Rhodus NL, Falace DA. Management of the dental patient with congestive heart failure. Gen Dent. 2002 May-Jun;50(3):260-5, quiz 266-7. PMID 12116514
- [Result] Blinder D, Manor Y, Shemesh J, Taicher S. Electrocardiographic changes in cardiac patients having dental extractions under a local anesthetic containing a vasopressor. J Oral Maxillofac Surg. 1998 Dec;56(12):1399-402; discussion 1402-3. doi: 10.1016/s0278-2391(98)90403-7. PMID 9846537
- [Result] Caceres MT, Ludovice AC, Brito FS, Darrieux FC, Neves RS, Scanavacca MI, Sosa EA, Hachul DT. Effect of local anesthetics with and without vasoconstrictor agent in patients with ventricular arrhythmias. Arq Bras Cardiol. 2008 Sep;91(3):128-33, 142-7. doi: 10.1590/s0066-782x2008001500002. English, Portuguese. PMID 18853053
- [Result] Dajani AS, Taubert KA, Wilson W, Bolger AF, Bayer A, Ferrieri P, Gewitz MH, Shulman ST, Nouri S, Newburger JW, Hutto C, Pallasch TJ, Gage TW, Levison ME, Peter G, Zuccaro G Jr. Prevention of bacterial endocarditis. Recommendations by the American Heart Association. Circulation. 1997 Jul 1;96(1):358-66. doi: 10.1161/01.cir.96.1.358. PMID 9236458